CLINICAL TRIAL: NCT00594685
Title: HIT Observational Thromboembolism Study (A TMH CTN Study)
Brief Title: Evaluating the Presence of Blood Clots in People With Heparin-Induced Thrombocytopenia (HIT) (The HOT Study)
Acronym: HOT
Status: Terminated | Type: Observational
Why Stopped: Low accrual rate
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 556; U01HL072299 (NIH); U01HL072299-01 (NIH); U01HL072268 (NIH); HL072033; HL072291; HL072289; HL072248; HL072191; HL072299; HL072305; HL072274; HL072028; HL072359; HL072072; HL072355; HL072283; HL072346; HL072331; HL072290
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Thrombocytopenia
Keywords: Heparin; Thromboembolism; Thrombosis
MeSH Terms: conditions — Thrombocytopenia; Thromboembolism; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and packed cells will be retained at Day 1 and Day 35 (+/- 7 days)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Isolated HIT: Hospitalized patients with isolated Heparin-Induced Thrombocytopenia (HIT), diagnosed by a fall in platelet count and a positive Platelet Factor 4 (PF4)-heparin Enzyme-Linked ImmunoSorbent Assay (ELISA) test

SUMMARY:
Heparin-induced thrombocytopenia (HIT), a condition characterized by low platelet levels and possible blood clots, occurs in a small number of people after treatment with the drug heparin. Some people with HIT may show symptoms of a blood clot at the time of HIT diagnosis, but in another form of HIT, known as isolated HIT, people do not show blood clot symptoms even though they might have a blood clot. This study will use ultrasound tests to evaluate the presence of blood clots at the time of an HIT diagnosis and in the following month.

DETAILED DESCRIPTION:
Heparin is a blood thinning medication that is often prescribed to treat or prevent blood clots. HIT is a life-threatening immune disorder that occurs in 1 to 3% of people who receive heparin. In this disorder, heparin does the opposite of what it is supposed to do: it promotes new blood clot formation, rather than preventing it. In people with HIT, the immune system triggers a response against heparin, leading to the destruction of platelets and a low platelet count, which is known as thrombocytopenia. Symptoms usually occur between 5 to 14 days after starting heparin therapy. Isolated HIT is a form of the condition that occurs when people have a low platelet count, but there is no sign of a blood clot, or thrombosis. Several small research studies have shown that at the time of isolated HIT diagnosis, between 15 to 50% of people actually have asymptomatic thrombosis, which means that they are not showing any signs of a blood clot, but in fact have one. In the month following HIT diagnosis, up to 50% of people experience symptomatic thrombosis, which means that they are showing signs of a blood clot. It is not currently known how to best treat isolated HIT and how to test for unrecognized blood clots. This study will use ultrasound imaging to evaluate the number of people who have asymptomatic thrombosis at the time of isolated HIT diagnosis and to determine the rate of symptomatic and asymptomatic thrombosis in the following month. The results of this study will assist researchers in assessing current approaches to treating isolated HIT and in designing new clinical trials. By exploring the use of non-invasive evaluation techniques in people with HIT, thrombosis research in HIT will move forward, similar to thrombosis research in other medical conditions.

This 29-day study will enroll hospital patients who have a diagnosis of HIT but show no signs of a blood clot at the time of HIT diagnosis. On Day 1, participants will undergo blood collection and an ultrasound. While participants are in the hospital, study researchers will review participants' medical records on a daily basis to collect data on current medications, medication compliance, symptoms, bleeding, thrombosis complications, and laboratory test results. Once participants leave the hospital, this data will be collected at least once a week through phone calls with the participant and/or the treating physician. On Day 29, participants will undergo a repeat ultrasound and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* In the 72 hours prior to study entry, participant has been diagnosed with "isolated HIT," as defined by an unexplained platelet count drop of over 50% that occurs after exposure to UFH (UnFractionated Heparin)/LMWH (Low Molecular Weight Heparin) at any time in the 4 to 14 days before the positive heparin-PF4 antibody test was sent(even if the person is no longer on UFH/LMWH)
* Currently hospitalized
* Available for study follow-up for at least 28 days after study entry
* No contraindications to ultrasound examination of upper and lower extremities
* For participants less than 7 years old, no contraindications to ultrasound examination of abdomen
* Participants are eligible whether or not they are receiving any therapy for isolated HIT

Exclusion Criteria:

* Documented new venous or arterial thrombosis while on heparin
* Pregnant
* Ongoing active bleeding (as determined by the site investigator)
* Currently using a extracorporeal membrane oxygenator, chronic veno-venous hemofiltration, left ventricular support device, intra-aortic balloon pump, or any other mechanical heart pump
* Coronary artery bypass surgery occured within 96 hours prior to the time when the positive HIT test was drawn

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients at participating clinical centers who have a diagnosis of isolated Heparin-Induced Thrombocytopenia (HIT), determined by a fall in platelet count after heparin treatment and a positive Platelet Factor 4 (PF4)-heparin Enzyme-Linked ImmunoSorbent Assay (ELISA) test
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Assmann, PhD, Principal Investigator — Carelon Research; Eliot C. Williams, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Kenneth D. Friedman, MD, Principal Investigator — Froedtert Hospital; David Kress, MD, Principal Investigator — St. Luke's Medical Center; Ronald Go, MD, Principal Investigator — Gunderson Clinic; Keith McCrae, MD, Principal Investigator — Case Western Reserve University; Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital; Jeff Zwicker, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Judith Lin, MD, Principal Investigator — Brigham and Women's Hospital; Thomas Ortel, MD, PhD, Principal Investigator — Duke University; Cassandra Josephson, MD, Principal Investigator — Emory University; Jodi Segal, MD, MPH, Principal Investigator — Johns Hopkins University; David Kuter, MD, Study Chair — Massachusetts General Hospital; Terry Gernsheimer, MD, Principal Investigator — University of Washington; Cindy Leissinger, MD, Principal Investigator — Tulane University; Thomas Raife, MD, Principal Investigator — University of Iowa; Ann Zimrin, MD, Principal Investigator — University of Maryland; Jeffrey McCullough, MD, Principal Investigator — University of Minnesota; Nigel Key, MB, MRCP, Principal Investigator — University of North Carolina; Ravindra Sarode, MD, Principal Investigator — University of Texas Southwestern Medical Center; Barbara Konkle, MD, Principal Investigator — University of Pennsylvania; Joseph Kiss, MD, Principal Investigator — University of Pittsburgh
Locations (21):
- United States (21):
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
  - Gunderson Lutheran Clinic, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isolated HIT
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Asymptomatic Thrombosis at the Time Isolated Heparin-Induced Thrombocytopenia (HIT) is Diagnosed, Determined by Four-limb Ultrasound
Description: The percentage of participants with asymptomatic thrombosis at the time isolated HIT is diagnosed as determined by four-limb ultrasound.
Time Frame: Measured at Day 1
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Percentage of participants | 20 [3 to 56]

2. Secondary Outcome: The Percentage of Participants With Asymptomatic Thrombosis 4 Weeks After the Diagnosis of Isolated HIT, Determined by Four-limb Ultrasound
Description: The percentage of participants with asymptomatic thrombosis 4 weeks after the diagnosis of isolated HIT, determined by four-limb ultrasound, and 95% exact binomial confidence interval.
Time Frame: Measured at Day 35 (+/- 7days)
Population: Four subjects had missing data for this endpoint (no ultrasound performed on end-of-study date) and are not included in this analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Isolated HIT
Number analyzed (Participants) | 6
Percentage of participants | 19 [0 to 64]

3. Secondary Outcome: The Number of Participants With Symptomatic Venous or Arterial Thromboembolism in the Month Following the Diagnosis of Isolated HIT
Description: There were two versions of the data collection form used in this study, and only the revised version collected information on whether the event was symptomatic.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: Two subjects did not have information on whether the event was symptomatic or asymptomatic. These two subjects were censored in the analysis.
Measure: Number; unit: Participants
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: The Number of Participants With Incidental Arterial and Venous Thromboembolism (i.e., a Clot Diagnosed by Radiographic Tests Done for Reasons Other Than to Diagnose or Rule Out a Thromboembolic Event)
Description: There were two versions of the data collection form used in this study, and only the revised form contained information on whether the event was incidental.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: Two subjects did not have information on whether the event was incidental. These subjects were censored in the analysis.
Measure: Number; unit: Participants
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: The Time to First Bleeding Event With Current Therapies for Isolated HIT
Description: The time to first bleeding event was analyzed using survival analysis.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days | 10.1 (2.2)

6. Secondary Outcome: Time Until Death From All Causes
Description: The time until death from all causes, in days, was determined using survival analysis.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: One subject was censored at the time that the study was terminated.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days | 12.2 (1.1)

7. Secondary Outcome: Time to Platelet Count Recovery
Description: The time to platelet recovery was defined as the time from the nadir platelet count observed in the five days after the positive HIT test was sent to observing a platelet count of 100K or greater. Survival analysis was used.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: One subject's nadir platelet count was > 100K, so that subject is not included in the analysis.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 9
Days | 2.9 (1.0)

8. Secondary Outcome: Number of Days That Medications Were Given to Participants at Participating Institutions
Description: Per the protocol, descriptive statistics on the types and durations of therapeutic approaches used will be presented.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Measure: Median (Full Range); unit: Days medication was given
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days medication was given
  Alteplase (Activase) - 1 subject | 11 [11 to 11]
  Argatroban - 4 subjects | 3.5 [3 to 4]
  Aspirin - 4 subjects | 36.5 [11 to 43]
  Clopidogrel (Plavix) - 2 subjects | 20.5 [4 to 37]
  Fondaparinux (Arixtra) - 3 subjects | 10 [6 to 11]
  Ibuprofen (Motrin, Advil) - 1 subject | 5 [5 to 5]
  Unfractionated Heparin - 3 subjects | 14 [2 to 18]
  Warfarin (Coumadin) - 5 subjects | 20 [1 to 40]

9. Secondary Outcome: Length of Hospital Stay
Description: The length of time between the date of HIT diagnosis and first hospital discharge was calculated. Subjects were censored at death. Survival analysis was used.
Time Frame: Measured upon hospital discharge
Population: Two subjects were known to be readmitted to the hospital after initially being discharged.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days | 10.4 (1.3)

10. Secondary Outcome: Length of Hospital Stay (With Deaths Not Censored)
Description: The length of time between the date of HIT diagnosis and first hospital discharge was calculated. Subjects were not censored at death. Survival analysis was used.
Time Frame: Measured upon hospital discharge
Population: Two subjects were known to be readmitted to the hospital after initially being discharged.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days | 10.1 (1.4)

11. Secondary Outcome: Relationship Between the Platelet Factor 4 (PF4)-Heparin Enzyme-Linked ImmunoSorbent Assay (ELISA) Test, the Serotonin-release Assay, and D-dimer Test Results
Description: Analysis not performed since central laboratory tests were not done.
Time Frame: Measured at Day 1
Population: Analysis not performed since central laboratory tests were not done.
Arm/Group | Isolated HIT
Number analyzed (Participants) | 0

12. Secondary Outcome: Relationship Between PF4-heparin ELISA Test, Serotonin-release Assay, and D-dimer Test Results and Thromboembolism
Description: Analysis not performed since central laboratory tests were not done.
Time Frame: Measured at Day 1 and within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: Analysis not performed since central laboratory tests were not done.
Arm/Group | Isolated HIT
Number analyzed (Participants) | 0

13. Post Hoc Outcome: Time to First Asymptomatic or Symptomatic Venous or Arterial Thromboembolism in the Month Following the Diagnosis of Isolated HIT
Description: Since two versions of the data collection form were used in this study, and only the revised version contained information on whether the event was asymptomatic or symptomatic, a post-hoc analysis was performed which included all thromboses, whether symptomatic, asymptomatic, or of unknown type. Survival analysis was used.
Time Frame: Measured within 35 days (+/- 7) after the diagnosis of isolated HIT
Measure: Mean (Standard Error); unit: Days
Arm/Group | Isolated HIT
Number analyzed (Participants) | 10
Days | 24.9 (2.8)

14. Secondary Outcome: Relationship Between the Presence of the Factor V Leiden Mutation or the Prothrombin 20210 Mutation and the Risk of Thrombosis
Description: Analysis not performed since central laboratory tests were not done.
Time Frame: Measured at Day 1 and within 35 days (+/- 7) after the diagnosis of isolated HIT
Population: Analysis not performed since central laboratory tests were not done.
Arm/Group | Isolated HIT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Within 35 days (+/- 7) after the diagnosis of isolated HIT
Description: The study will collect data on thromboses and on bleeding events, the two types of adverse events most commonly associated with HIT and its treatment. Data will also be collected on all serious adverse events that are attributed as being possibly, probably, or definitely related to involvement in the study.
Arm/Group | Isolated HIT
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isolated HIT (N=10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study due to low enrollment. Due to the early termination, the central laboratory tests necessary for analyzing outcomes 11, 12, and 13 were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No